



# Clinical and Radiographic Evaluation of Delayed Implant Placement Following Socket Preservation with Injectable Alloplastic Bone Graft: A Randomized Controlled Study.

A Thesis Protocol
Submitted for partial fulfillment of the requirements of the
Master degree in dental science
In

# Oral and Maxillofacial Surgery

Research code: HE 11

Submitted By

#### **Ahmed Rawhy Mounir Saleh**

M.U.S Mansoura University 2019 Dentist at The Egyptian ministry of health ,2021

#### **Supervisors**:

| Title | Name | Job Title | University | Signature |
|-------|------------|----------------------|------------|-----------|
| Prof. | Mohamed | Professor of Oral | Suez Canal | |
| | Ahmed | and Maxillofacial | University | |
| | Elsholkamy | Surgery | | |
| | | Department, Faculty | | |
| | | of Dentistry | | |
| Dr. | Mohamed | Lecturer in oral and | Suez Canal | |
| | Nageh Gad | maxillofacial | University | |
| | ElHak | Surgery, Faculty of | | |
| | | Dentistr | | |

Faculty of Dentistry

**Suez Canal University** 

2025



# "Thesis Research Protocol"

| Student Name: | Ahmed Rawhy Mounir Saleh | | Student | 29605191301178 |
|---|---|---|---|---|
| | | | ID: | |
| Submission | 4/29/2025 | | | |
| Date: | | | | |
| Degree: | ☐ PH.D. | | | |
| Department: | Suez Canal Un | iversity | | |
| | Clinical and Radiographic Evaluation of | | | |
| Thesis Title in | Delayed Implant Placement Following Socket | | | |
| English: | Preservation with Injectable Alloplastic Bone | | | |
| | Graft. A Rar | ndomized | Controlle | ed Trial. |
| Thesis Title in | ة بعد حفظ تجويف | سات المتأخر | بي لوضع الغر | التقييم السريري والشعاء |
| Thesis Title in Arabic: | ـ دراسة عشوائية | ي قابل للحقن | ىي غير عضو: | السن باستخدام طعم عظه |
| Alubici | | | | محكمة |



#### 1. Abstract

Introduction: Tooth extraction leads to alveolar ridge resorption which can compromise future implant placement. Socket preservation using alloplastic bone grafts may help maintain ridge dimensions and allow for predictable delayed implant placement. Injectable alloplastic bone substitutes have gained attention due to their ease of handling and osteoconductive properties. Aim: To evaluate the clinical and radiographic outcomes of delayed implant placement after socket preservation using injectable alloplastic bone graft. Methodology: Twenty Implants will be placed in 20 patients that have previously extracted a lower posterior tooth, . Group (1): patients without socket preservation after extraction . Group (2): patients with socket preservation after extraction . Clinical outcomes including soft tissue healing, implant stability, and postoperative complications will be assessed. Radiographic evaluation using CBCT will be made before implant placement, and after 6 months to measure changes in ridge width and height.



## 2. Introduction and Background

Tooth extraction is often associated with significant remodeling of the alveolar ridge. This natural biological process results in resorption of the alveolar bone, with the greatest volume of bone loss occurring within the first 3–6 months following extraction .Studies have shown that horizontal bone loss can reach up to 50% in width and 60% in height during this period (Van der Weijden et al., 2009).

This resorptive process is not only a physiological consequence of tooth loss but also a critical challenge for the prosthetically-driven placement of dental implants .Alveolar ridge preservation (ARP) techniques have been developed to mitigate this bone loss by preserving the ridge volume immediately following extraction .ARP commonly involves the placement of bone graft materials into the extraction socket, often with or without a barrier membrane, to support new bone formation and maintain soft tissue contours (Avila-Ortiz et al., 2014).

Multiple types of bone grafts have been introduced for this purpose, including autografts, allografts, xenografts, and alloplastic materials, each with distinct biological and handling properties .Alloplastic grafts, which are synthetic in nature, offer several advantages such as biocompatibility, lack of disease transmission risk, and ease of manipulation. Among these, injectable alloplastic bone substitutes have gained increasing popularity due to their moldability, minimally invasive application, and ability to conform precisely to the defect morphology (Mangano et al., 2013).

These materials generally consist of calcium phosphate or sulfate compounds and function primarily through osteoconduction, providing a scaffold for bone in-growth (Jensen et al., 2006).

Their injectable nature allows for easy delivery into the socket without the need for extensive surgical manipulation, thus reducing chair time and improving patient comfort. While immediate implant placement is sometimes employed in ideal conditions (i.e., intact bony walls, absence



of infection), it is not always feasible or advisable. Clinical situations involving thin biotypes, bone deficiencies, or aesthetic demands often necessitate a delayed implant placement protocol to allow for adequate tissue healing and graft maturation (Chen & Buser, 2009).

In such scenarios, prior socket preservation may significantly influence the quality and quantity of bone available at the time of implant placement.

Several clinical trials and systematic reviews have demonstrated the effectiveness of socket preservation procedures in reducing post-extraction dimensional changes and enhancing the conditions for implant placement (Mardas et al., 2015; Vignoletti et al., 2012).

However, the specific role of injectable alloplastic materials in socket preservation—particularly in terms of long-term clinical and radiographic outcomes—remains underexplored. Additionally, there is limited evidence regarding the bone quality they produce in healed sites and their influence on primary implant stability. Cone beam computed tomography (CBCT) has become the gold standard for evaluating dimensional bone changes due to its high accuracy and low radiation dose. It allows for detailed 3D assessment of bone volume, ridge width, height, and density (Bornstein et al., 2014).

Upon search of literature, up-to knowledge there are insufficient studies assessing delayed implant placement following socket preservation with injectable bone graft, hence, the aim of the present study.

# 3. Research Q (RQ):

In patients that require delayed implant in posterior mandible, what is the effect of delayed implant placement following socket preservation with Injectable bone graft? Clinically regarding implant stability, soft tissue healing and postoperative pain. As well as radiographically regarding horizontal and vertical dimensional changes in the alveolar ridge?



#### 4. Research Hypothesis, Aim, Objectives & Expected Outcomes

#### a. Hypothesis

Null Hypothesis (H<sub>0</sub>):

There is no significant difference in the effect of delayed implant placement following socket preservation in comparison to implant placement without socket preservation.

Alternative Hypothesis (H<sub>1</sub>):

There is a significant difference in the behavior of delayed implant placement following socket preservation in comparison to implant placement without socket preservation.

#### b. Aim

To evaluate the clinical and radiographic outcomes of delayed implant placement after socket preservation using injectable alloplastic bone graft.

## c. Objectives

Clinical parameters:

- 1)Measure implant stability at the time of placement and after osseointegration using OSTELL .(immediately after implant placement and 6 month after implant placement)
- 2)Assess soft tissue healing and wound dehiscence by visual inspection (one week after the surgery)
- 3)Monitor postoperative pain by VAS and swelling through visual inspection and palpation .(Day 1, Day 3 ,and Day 7 postoperatively)
- 4)Record any complications (infection, graft exposure, etc.) by visual inspection .(afte one week)

Radiographic parameters:

1)Measure horizontal and vertical dimensional changes in the alveolar



ridge after 6 months using CBCT.

2)Evaluate the radiographic bone density at the grafted site (after 6 months)

## d. Expected Outcomes

Socket preservation using injectable alloplastic bone graft may reduce alveolar ridge resorption, enhance bone quality at the implant site, and facilitate optimal implant placement.



# 5. Research Design and Methods

#### 1- Materials:

| item | Туре | Manufacturer |
|---|---|---|
| Dental implant | Titanium | SGS Turkey |
| Local anesthetic | Articaine 4% with epinephrine 1:100,000 | Alexadricaine |
| Sutures | 4-0 or 5-0 resorbable/non-resorbable sutures | Asset suture |

#### 2- Methods

#### A -Study Design:

Controlled clinical study, randomization has been done for the patients before extraction and socket preservation using http://www.randomizer.org

#### **B** – Study Settings:

Outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Suez Canal University.

## **C-Study population:**

20 patients requiring delayed implant placement in posterior mandibular region, the patients will be divided into 2 equal groups (n = 10 per group).

# 1-Patient selection and eligibility criteria

Inclusion criteria: (Lin et al., 2019, Mandelli et al., 2019)

- Patient aged between 40 and 60 years
- General good health.
- Volunteer subjects have to voluntarily sign an informed consent.
- Patient Indicated for single implant placement in lower posterior area.



#### Inclusion criteria for patients in group I

• Patient with a previously extracted lower posterior tooth and the socket was preserved with injectable bone graft.

#### Exclusion criteria: (Lin et al., 2019, Mandelli et al., 2019)

- Patient with systemic disease affection bone metabolism.
- Patients with contraindication to surgical treatment.
- Patients with uncontrolled medical conditions.

#### 2-Patient Grouping:

#### **Group I (Test Group):**

Including 10 patients with extracted mandibular posterior tooth who undergone socket preservation with Injectable alloplastic bone graft.

## **Group II (Control Group):**

Including 10 patient with extracted mandibular posterior tooth and left for natural healing.

# D -Methodology

# Pre-operative assessment.

Clinical assessment will also include evaluation of soft tissue quality, keratinized gingiva, and occlusal considerations to ensure proper implant planning (Bornstein et al., 2014).

# Radiographic assessment

Before implant placement, patients will undergo radiographic evaluation, including cone-beam computed tomography (CBCT) to assess alveolar ridge dimensions, bone density, and anatomical structures such inferior alveolar nerve. At 4 months post-extraction, prior to implant placement (baseline)



#### **CBCT** Equipment Specifications:

- Device: Scanora 3D by Soredex (Tuusula, Finland)
   Specifications
- Imaging type: CBCT with optional high-resolution 2D panoramic
- Fields of View (FOV):  $60 \times 60$  mm,  $75 \times 100$  mm,  $75 \times 145$  mm, optional XL up to  $130 \times 145$  mm
- Voxel size: 0.4 mm
- Scan time: 8–30 sec (effective exposure 2–7.5 sec)
- X-ray tube: 60–90 kV, 1.0–8.0 mA, fixed anode
- Focal spot: 0.5 mm (IEC 60336)
- Detector: Flat panel (CBCT), CCD (panoramic)
- Features: AutoSwitch between CBCT and panoramic
- Dimensions: 1973 × 1600 × 1400 mm

Patients will be scanned in a seated upright position with a rigid head support to minimize motion artifacts.

#### **Surgical Protocol:**

The dental implant placement will be performed under strict aseptic conditions and following standard surgical protocol for delayed implantation. The procedure will take place approximately 4 months following tooth extraction and socket preservation for patient in both groups. (Peitsinis et al., 2025; ITI, 2018)

# 1. Preoperative Preparation (Esposito et al., 2023):

- Patient will rinse with 0.12% chlorhexidine gluconate mouthwash for 1 minute.
  - Extraoral skin will be disinfected with povidone-iodine.
- Local anesthesia will be administered using 4% Articaine with 1:100,000 epinephrine via infiltration or nerve block as needed.

# 2. Surgical Access(Misch, 2021):

- A mid-crestal incision will be made in the edentulous ridge using a scalpel blade no.15.
  - Two small vertical releasing incisions may be added to ensure



adequate access, depending on tissue quality.

• A full-thickness mucoperiosteal flap will be reflected to expose the underlying alveolar bone.

#### 3. Osteotomy Preparation(Misch, 2021):

Standard clinical guidelines will guide the implant position (based on CBCT).

- A round bur will be used to mark the implant site. (Misch, 2021)
- Sequential drills of increasing diameter (pilot drill, twist drills) will be used at low speed (800–1200 rpm) under copious sterile saline irrigation to prepare the osteotomy to the desired depth and diameter according to the implant system used.
- Direction indicators or paralleling pins may be inserted intermittently to verify angulation and position.

#### 4. Implant Insertion(Misch, 2021):

- The titanium dental implant will be inserted into the prepared site using either a hand ratchet or implant motor at controlled torque (typically 30–45 Ncm).
- Primary stability will be assessed using resonance frequency analysis (e.g., Osstell ISQ).
  - A healing abutment or cover screw will be placed.
- Flap will be repositioned and sutured using 4-0 or 5-0 non-resorbable or resorbable sutures using interrupted or horizontal mattress technique. (Misch, 2021)

# 5. Postoperative Instructions and Medications (Esposito et al., 2023)

- The patient will be instructed to maintain strict oral hygiene and avoid brushing near the surgical site for 7 days.
- Chlorhexidine mouth rinse 0.12% twice daily for 10 days will be prescribed.
- Analgesics (e.g., ibuprofen 600 mg every 8 hours as needed) and antibiotics (e.g., amoxicillin/clavulanic acid 1 g twice daily for 5 days) will be administered.



#### 6. **Follow-up (ITI, 2018):**

- Sutures will be removed after 7–10 days. (Misch, 2021)
- Healing will be monitored clinically and radiographically.
- Osseointegration will be reassessed after 3 months, and if satisfactory, prosthetic loading will be initiated.
- Abutment will be placed and impression will be taken to get the final restoration loading.

#### **Post-operative Assessment**

#### **A-Clinical Evaluations**

**1-Implant Stability** will be assessed using a non-invasive method based on resonance frequency analysis (RFA) utilizing the Osstell ISQ® device. This technique provides a quantitative measure of the implant's mechanical stability in bone and is highly predictive of osseointegration success (Meredith, 1998; Ostman et al., 2006).

After implant insertion, a smart peg compatible with the implant system will be attached to the implant fixture using the manufacturer's torque recommendation (approximately 4–6 Ncm). The Osstell probe will then be positioned near the peg without contact to transmit magnetic pulses.

Measurements will be taken in two directions (buccolingual and mesiodistal), and the mean Implant Stability Quotient (ISQ) will be calculated. The ISQ scale ranges from 1 to 100, with values above 65 generally indicating high primary stability suitable for early or immediate loading (Sennerby & Meredith, 2008).

Stability will be measured at the time of implant placement and again after a healing period of 6 months to assess secondary (biological) stability.

**2-Postoperative pain** will be evaluated using the Visual Analog Scale (VAS), a widely accepted and validated method for measuring subjective pain perception in clinical dental studies. The VAS is a 10-centimeter horizontal line with endpoints defined as "0" (no pain) and "10" (worst



imaginable pain). Patients will be instructed to mark the line at the point that best represents their pain intensity at predefined intervals: Day 1, Day 3, and Day 7 postoperatively. (Alghamdi et al., 2023).

- **3-Soft Tissue Healing**: Careful examination of the surgical site to assess epithelialization, and detection of any wound dehiscence or delayed soft tissue healing one week after surgery (Buser et al., 2017).
- **4. Complication Monitoring**: Recording of any complications such as infection, graft exposure, hematoma, suture dehiscence, or early implant mobility. These events will be documented systematically for subsequent analysis (Esposito et al., 2013).

#### **B-Radiographic Assessment**

Radiographic evaluation will be performed using Cone Beam Computed Tomography (CBCT) to assess dimensional and qualitative changes in the alveolar ridge at different stages of the study. CBCT provides high-resolution three-dimensional imaging and has become the gold standard for quantitative bone analysis in implant dentistry (Gonzalez-Garcia et al., 2023). All images will be evaluated using dedicated on demand for consistent calibration.

Scans will be taken at the following time points:

• 6 months post-implantation to assess bone remodeling around the implant

Parameters to be assessed include (Alssum et al., 2025; Gong et al., 2024):

- 1) Marginal bone level changes.
- 2) Vertical ridge height (buccal and lingual/palatal aspects)
- 3) Bone density around the implant (in Hounsfield Units)
- 4) Buccal plate thickness.



# 6. Statistical plan

# a) Sample size calculation:

#### will be two-tailed (Chan Y, 2003).

#### Sample size calculation:

The sample size for this study was calculated according to Chan, 2003 and used the following equation: (Chan Y, 2003)

$$N = \frac{(\mathbf{Z}\alpha)^2 * (S)^2}{(d)^2}$$

N = Total sample size,

 $Z\alpha$ = Is Standard normal variate and its equal to 1.96 at P< 0.05,

SD = Standard deviation of variable,

d = Absolute error or precision

| Zα | SD | D |
|------|-----|---|
| 1.96 | 4.6 | 2 |

$$N = \frac{(1.96)^2 * (4.6)^2}{(2)^2} = 20.3 \approx 20 \text{ implants}$$

The total sample size calculations revealed that the sample size should be 20 samples



will be divided equally as follows:

| Groups | Descriptive | Samples |
|---------|----------------------------------------|---------|
| Group A | Implants in Sockets preserved with IBS | 10 |
| Group B | Implants in Empty socket | 10 |

This sample size is in agreement with previous study that test in similar subject

#### (Mandelli et al., 2019)

#### **Statistical analysis:**

Data will be coded and entered using the statistical package SPSS version 22. Data will be summarized using mean and standard deviation. Data will be explored for normality using the Kolmogorov-Smirnov test. Comparisons between both groups for normally distributed data will be done using a t-test. P value less than or equal to 0.05 will be considered statistically significant.

# 7. Ethics consideration

The present research will be conducted after the approval of the Research Ethics Committee (REC) of the Faculty of Dentistry, Suez Canal University. It will be conducted on twenty patients who meet the inclusion criteria specified in the study. Ethical considerations regarding patient well-being, safety, and confidentiality will be undertaken by the researcher.

An informed written consent will be signed by all subjects/patients before commencing the study. The consent will explain the clinical examinations, procedures, potential risks, benefits, and the follow-up



required for participation in the study. explain the clinical examinations, procedures, potential risks, benefits, and the follow-up required for participation in the study.

#### 8. Time Plan

 $\textbf{Starting} \ \textbf{After approval of the Ethical Committee and faculty council.} \ \textbf{Ending} : \textbf{12 Months}$ 

#### **Include Grant Chart as following example:**

| Activity/Month | 1 | 2 | 3 | 4 | 5 | 9 | 7 | 8 | 6 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Ethical Approval & Preparation | ⊠ | | | | | | | | | | | | | | | | | | | | | | | |
| Patient Selection & Consent | | × | | | | | | | | | | | | | | | | | | | | | | |
| Implant Placement | | | | × | × | | | | | | | | | | | | | | | | | | | |
| Final Evaluations | | | | | | × | × | × | × | × | ☒ | × | | | | | | | | | | | | |
| (Clinical&CBCT) | | | | | | | | | | | | | | | | | | | | | | | | |
| Statistical Analysis | | | | | | | | | | | | | M | | | | | | | | | | | |
| Writing & Submission. | | | | | | | | | | | | | | × | | | | | | | | | | |

# 9. Research Estimated Budget in Egyptian Pound

| Radiographs | drugs/<br>Lab chemicals | Lab-investigations<br>Software | Material | Others<br>(mention) | Publications | Total |
|---|---|---|---|---|---|---|
| CBCT | Antibiotics,<br>analgesics,<br>anti-<br>inflammatory<br>Drugs | Implant systems 20<br>implant | Lancet#15,<br>Suture silk<br>, Local<br>anesthesia,<br>Saline | | | |
| 10000 | 1500 | 48000 | 2000 | | 2000 | 63500 |



#### 10. References

- Alghamdi, H.S., AlShahrani, M.A., AlAmri, M.D. and Alfayez, M., 2023. Evaluation of postoperative pain following different dental implant protocols using visual analog scale: A clinical observational study. Journal of Oral and Maxillofacial Surgery, Medicine, and Pathology, 35(1), pp.25–30.
- Alssum, L., Alhazmi, A., Alanazi, A., Alruwaili, M., Alsughayyir, M., Alotaibi, T., Alanazi, M. and Alqahtani, M., 2025. Clinical and radiographic evaluation of bone profile and soft tissue parameters around implants placed in preserved sockets: a prospective study. Journal of Clinical Medicine, 14(2), p.367.
- Avila-Ortiz, G., Elangovan, S., Kramer, K.W.O., Blanchette, D. and Dawson, D.V., 2014. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. Journal of Dental Research, 93(10), pp.950–958.
- Bornstein, M.M., Halbritter, S., Harnisch, H., Weber, H.P. and Buser, D., 2014. Cone beam computed tomography for diagnosis and treatment planning in implant dentistry: a systematic review. International Journal of Oral and Maxillofacial Implants, 29(Suppl), pp.125–139.
- Buser, D., Sennerby, L. and De Bruyn, H., 2017. Modern implant dentistry based on osseointegration: 50 years of progress, current trends and open questions. Periodontology 2000, 73(1), pp.7–21.
- Chan, H.L., 2003. The significance of alveolar ridge dimensions in implant dentistry. Clinical Oral Implants Research, 14(2), pp.137–148.



- Chappuis, V., Araújo, M.G. and Buser, D., 2017. Clinical relevance of dimensional bone and soft tissue alterations post-extraction in esthetic sites. Periodontology 2000, 73(1), pp.73–83.
- Chen, S.T. and Buser, D., 2009. Clinical and esthetic outcomes of implants placed in postextraction sites. International Journal of Oral and Maxillofacial Implants, 24(Suppl), pp.186–217.
- Esposito, M., Grusovin, M.G. and Worthington, H.V., 2013. Interventions for replacing missing teeth: antibiotics at dental implant placement to prevent complications. Cochrane Database of Systematic Reviews, (7), CD004152.
- Esposito, M., Cannizzaro, G., Barausse, C., Felice, P. and Buti, J., 2023. Immediate and delayed implant placement: a systematic review and meta-analysis. European Journal of Oral Implantology, 16(2), pp.99–116.
- Gong, Z., Xu, H., Luo, Z., Chen, H., Huang, X. and He, F., 2024. Influence of bone conditions on the accuracy of implant placement using static computer-assisted surgery: A CBCT study. Journal of Clinical Medicine, 13(10), p.2804.
- Gonzalez-Garcia, R., Monje, A. and Hernández-Alfaro, F., 2023. Role of cone-beam computed tomography in dental implantology: a critical review of current evidence and future perspectives. Clinical Oral Implants Research, 34(2), pp.190–204.
- International Team for Implantology (ITI), 2018. ITI Treatment Guide. Volume 4: Immediate Implant Placement. Berlin: Quintessence Publishing.
- Jensen, S.S., Broggini, N., Hjørting-Hansen, E., Schenk, R. and Buser, D., 2006. Bone healing and graft resorption of autograft, anorganic bovine bone and β-tricalcium phosphate. Clinical Oral Implants Research, 17(3), pp.237–243.
- Lin, G.H., Lim, G., Chan, H.L., Giannobile, W.V. and Wang, H.L., 2019. Recombinant human bone morphogenetic protein 2 outcomes for alveolar ridge preservation: a systematic review and meta-analysis. Clinical Oral Implants Research, 30(8), pp.773–782.
- Mandelli, L., Rossi, G. and Bianchi, F., 2019. Bone regeneration with injectable alloplastic materials: a clinical and radiographic study. Journal of Oral Implantology, 45(2), pp.123–130.
- Mangano, C., Piattelli, A., Mangano, F., Mangano, R., Mangano, A. and Iezzi, G., 2013. Prospective clinical evaluation of 201 direct laser metal forming implants: results from a 1-year multicenter study. Lasers in Medical Science, 28(2), pp.641–648.



- Mardas, N., Trullenque-Eriksson, A., MacBeth, N. and Donos, N., 2015. Does ridge preservation following tooth extraction improve implant treatment outcomes? A systematic review. Clinical Oral Implants Research, 26(Suppl 11), pp.180–201.
- Meredith, N., 1998. Assessment of implant stability as a prognostic determinant. International Journal of Prosthodontics, 11(5), pp.491–501.
- Misch, C.E., 1999. Contemporary Implant Dentistry. 2<sup>nd</sup> edn. St. Louis: Mosby Elsevier.
- Misch, C.E., 2021. Contemporary Implant Dentistry. 4<sup>th</sup> edn. St. Louis: Mosby Elsevier.
- Ostman, P.O., Hellman, M. and Sennerby, L., 2006. Direct implant loading in the edentulous maxilla using a bone density—adapted surgical protocol and primary implant stability criteria for inclusion. Clinical Implant Dentistry and Related Research, 8(4), pp.173–182.
- Peitsinis, A., Kanatas, A. and Greenwood, M., 2025. Clinical decision-making in immediate versus delayed implant placement: a systematic review. Journal of Oral Rehabilitation, 52(3), pp.321–334.
- Sennerby, L. and Meredith, N., 2008. Implant stability measurements using resonance frequency analysis: biological and biomechanical aspects and clinical implications. Periodontology 2000, 47(1), pp.51–66.
- Troiano, G., Zhurakivska, K., Lo Muzio, L. and Laino, L., 2017. Combination of platelet-rich fibrin and bone grafts in alveolar ridge preservation: a systematic review. Journal of Oral and Maxillofacial Surgery, 75(7), pp.1501–1511.
- Van der Weijden, F., Dell'Acqua, F. and Slot, D.E., 2009. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. Journal of Clinical Periodontology, 36(12), pp.1048–1058.
- Vignoletti, F., Matesanz, P., Rodrigo, D., Figuero, E., Martín, C. and Sanz, M., 2012. Surgical protocols for ridge preservation after tooth extraction. A systematic review. Clinical Oral Implants Research, 23(Suppl 5), pp.22–38.



# 11. Appendices

(Questionnaire / Consent form)

# Faculty of Dentistry Research Ethics Committee (REC)

## **Investigator Application Form**

1- Name of researcher: Ahmed Rawhy Mounir Saleh

2- Name of Department: Oral and Maxillofacial Surgery

3- Address of researcher: Ibrahimia sharqia.

a- Email: ahmedrawhi96@gmail.com

b- Phone number: 01022552382

4- Name (s) of Co-investigator (s):

Prof. Dr. Mohamed Ahmed Elsholkamy

Dr. MohamedNageh Gad El Hak

5- Grade of protocol:



```
*M.D.Sc. (✓)
   *Ph.D. ( )
   *Doctorate degree (D.D.Sc)
   *Other()
   *Domestic ()
   *Multi-Centre within Egypt()
   *International()
6-Title of the research Clinical and Radiographic Evaluation of
Delayed Implant Placement Following Socket Preservation with
Injectable Alloplastic Bone Graft.
7-Type of the research:
  *Drug trial ()
  *Surgical technique (\checkmark)
  *Investigative technique ()
  *Devise study ()
  *Survey study ()
  *Blood sampling ()
  *Review Of old records ()
  8 - Subjects of research
   * Children (< 18 years): ( )
                                 *Adults (>18 years) : (√)
  9-Request is being made to waive(give-up) informed consent:
         Yes (√) No ( )
  10-The research is for the good of society: yes (\checkmark)no ()
  11-Study design:
                       I: ( ) II: ( ). III: ( )
  a-Phase type
  b-Randomization:
                        Yes: ( √ ) No: ( )
```



c-Placebo: Yes: ( ) No: ( )
d-Genetic sampling: Yes: ( ) No: ( )
e-Other: Yes: () No: ( )

12- Facilities for the research are available: yes (✓) No: ( )

#### 13-List the risks of the study:

- 1. Infection at the surgical site.
- 2. Pain or swelling during the healing phase.
- 3. Graft failure or insufficient bone regeneration.
- 4. Allergic reaction or sensitivity to the graft material (rare).
- 5. Implant failure due to poor osseointegration (in rare cases).
- 14-List the potential benefits, if any, to the subjects:
- 1. Preservation of bone volume after tooth extraction, reducing the risk of future bone loss.
- 2. Improved implant stability due to better bone quality.
- 3. More predictable implant placement with proper bone dimensions.
- 4. Enhanced aesthetic outcomes, especially in visible areas.
- 5. Minimally invasive handling of the graft material (injectable).
- 6. Reduced need for additional bone grafting procedures later.
- 7. Better healing of soft tissues due to ridge preservation.

15-Are the risks reasonable to the potential benefits to the subjects, if any, or to the knowledge to be gained? Yes:  $(\checkmark)$ 



| No: ( ) | |
|---|---|
| 16-Privacy and confidentiality of subjects are assur | red Yes: ( <u>√</u> ) No: ( ) |
| 17-The subject of the research could quit at any time | without penalty |
| or loss of any benefits to which they would otherwis | e be entitled: |
| Yes: ( <b>✓</b> ) No: ( ) | |
| 18- All surgeries will done under supervision of prof | essors |
| Signature of the principal investigator: | Date: |